CLINICAL TRIAL: NCT01025102
Title: Phase III Study of the Addition of Sufentanil to Interscalene Block in Shoulder Surgery
Brief Title: The Addition of Sufentanil Interscalene Block in Shoulder Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bent Gymoese Jorgensen (Other)
Responsible Party: Sponsor-Investigator, Bent Gymoese Jorgensen, MD, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: gymoese007
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Postoperative Pain; Shoulder Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naropin 0.1% (Experimental)
  Interventions: Drug: Naropin 0.1% cum sufentanil

INTERVENTIONS:
Drug: Naropin 0.1% cum sufentanil — 20ml of Naropin 0.1% cum sufentanil 1mikrog per ml
  Other Names: Local analgetic; Ropivacain

SUMMARY:
The purpose of this study is to compare the effects and side effects of interscale block performed with Naropin 0.1% cum sufentanil or Naropin 0.1% in shoulder surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare the duration of postoperative analgesia and supplemental opioid consumption and side effects of interscale block performed with Naropin 0.1% cum sufentanil or Naropin 0.1% in shoulder surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80
* Shoulder surgery performed under interscalene block and general anesthesia

Exclusion Criteria:

* Contraindication of interscalene block
* Severe chronic obstructive lung disease
* Non-cooperative patient
* Intolerance to opioids
* Pregnancy
* Rheumatoid arthritis and diabetes with peripheral polyneuropathy
* Chronic pain or daily opioid intake

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to experience of moderate to severe postoperative pain | On day of surgery and 1., 2. and 3. postop. day

SECONDARY OUTCOMES:
Side effects | On day of surgery and 1., 2. and. 3. postop. day

CONTACTS AND LOCATIONS:
Overall Officials: Bent G Jørgensen, MD, Principal Investigator — Anesthetic Clinic, Frederiksberg University Hospital
Locations (1):
- Anesthetic Clinic, Frederiksberg University Hospital, Frederiksberg, Frederiksberg, Denmark